CLINICAL TRIAL: NCT07376174
Title: A Multicenter Retrospective Cohort Study Protocol on the Prognostic Impact of HER2 Expression in Non-Metastatic HER2-Positive Breast Cancer Treated With Dual HER2-Targeted Therapy
Brief Title: The Prognostic Impact of HER2 Expression in Non-Metastatic HER2-Positive Breast Cancer Treated With Dual HER2-Targeted Therapy
Status: Recruiting | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Fangchao Zheng, MD, Clinical associate professor, Shandong Cancer Hospital and Institute
Other Study IDs: SDTHEC202601024
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HER2/CEP17 Ratio
Keywords: HER2/CEP17 ratio; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2 FISH ultra: HER2/CEP17 FISH ratio in HER2-positive non-metastatic breast cancer
- HER2 FISH normal: HER2/CEP17 FISH ratio in HER2-positive non-metastatic breast cancer

SUMMARY:
Previous studies suggest that among patients receiving trastuzumab monotherapy, a HER2/CEP17 ratio >7.0 (ultra-high expression) is associated with poorer disease-free survival (DFS). Dual-target therapy (trastuzumab + pertuzumab) has become the standard treatment for high-risk HER2-positive breast cancer; however, whether it can predict outcomes in patients with ultra-high HER2 expression remains unsupported by clinical data. To analyze the clinicopathological characteristics and prognostic relationship between the HER2 ultra-high expression group and the normal expression group in non-metastatic HER2-positive breast cancer patients who received dual-target therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Pathologically confirmed primary breast cancer, clinical stage I-III (AJCC 8th Edition).
3. HER2-positive status confirmed by FISH testing (per ASCO/CAP guidelines) with available HER2/CEP17 ratio.
4. Received at least one dose of dual-target therapy (trastuzumab combined with pertuzumab) in the adjuvant or neoadjuvant setting.
5. Underwent curative-intent surgery (mastectomy or breast-conserving surgery).

Exclusion Criteria:

1. Presence of distant metastasis (Stage IV) or contralateral breast cancer at initial diagnosis.
2. Previous anti-HER2 targeted therapy prior to dual-target treatment.
3. Missing key clinical data (e.g., HER2 FISH results, treatment regimen, surgery date).
4. Carcinoma in situ or occult breast cancer, non-primary breast cancer, or concurrent other malignancies.
5. Loss to follow-up or follow-up duration <3 months (unless recurrence or death occurred within this period).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive patients with breast cancer were enrolled between January 2020 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival based on HER2/CEP17 ratio | From the date of pathological diagnosis to event with follow-up duration ≥3 months (unless recurrence or death occurred within 3 month).
  Defined as the period from the date of pathological diagnosis until the date of the first relapse, appearance of non-breast primary cancer, death with no signs or symptoms of recurrence or metast, or the last recorded follow-up ,whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Jinan, Shandong, China